CLINICAL TRIAL: NCT03111784
Title: Effect of Fish Consumption on Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern University, Sri Lanka (Other)
Collaborators: Ministry of Health, Sri Lanka (Other Government)
Responsible Party: Principal Investigator, Chandravathany Devadawson, Senior Lecturer, Eastern University, Sri Lanka
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EasternU
Record Dates: First submitted 2017-04-08; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Fish Consumers
Keywords: Fish Consumption, Fatty acid composition, Lipid Profile, Tocopherol, Sociodemographics

STUDY DESIGN:
Intervention Model Description: Quasi Experimental / non-randomised trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fish consumption and lipid profiles

SUMMARY:
IConsumption of fish provides a vital contribution to the survival and health of a significant portion of the world's population. Lipids in fish foods consist mainly of long-chain polyunsaturated fatty acids (PUFAs) such as eicosapentaenic acid (EPA, C20:5n-3) and docosahexaenoic acid (DHA C22:6n-3) which belongs to the physiologically important group of n-3 fatty acids. The increase of unsaturated fatty acids, along with the reduction of saturated fats, supports the lowering of blood cholesterol in humans and causes a positive impact on human nutrition. Polyunsaturated fatty acids (omega-3 fatty acids) plays a role in preventing heart disease and has anti-inflammatory and anti-thrombosis effects and these fatty acids cannot be synthesized and they must be obtained through diet. These nutritional benefits of fish consumption is mainly attributed to the effect of omega-3 polyunsaturated fatty acids , which are thought to have several potential cardio protective actions. This research is focused mainly identify highly consumed food fishes available in Batticaloa district( fresh, lagoon and sea water ) and their consumption pattern (cooking methods) of local community and by cardiovascular patients (CV) . Secondly Omega-3- Polyunsaturated fatty acid (PUFA) and tocopherol content (Vit E) in the fresh fish and dried or smoked fish of the highly consumed food fishes would be assessed and the relationship between fish consumption and its PUFA and Vit E content would be known. Also research will focus how lifestyle, socio-demographic factors' influences on the Cardiovascular diseases among community.

DETAILED DESCRIPTION:
1. Introduction

   Consumption of fish provides a vital contribution to the survival and health of a significant portion of the world's population. Lipids in fish foods consist mainly of long-chain polyunsaturated fatty acids (PUFAs) such as eicosapentaenic acid (EPA, C20:5n-3) and docosahexaenoic acid (DHA C22:6n-3) which belongs to the physiologically important group of n-3 fatty acids. The increase of unsaturated fatty acids, along with the reduction of saturated fats, supports the lowering of blood cholesterol in humans and causes a positive impact on human nutrition. Polyunsaturated fatty acids (omega-3 fatty acids) plays a role in preventing heart disease and has anti-inflammatory and anti-thrombosis effects and these fatty acids cannot be synthesized and they must be obtained through diet. These nutritional benefits of fish consumption is mainly attributed to the effect of omega-3 polyunsaturated fatty acids , which are thought to have several potential cardio protective actions. This research is focused mainly identify highly consumed food fishes available in Batticaloa district( fresh, lagoon and sea water ) and their consumption pattern (cooking methods) of local community and by cardiovascular patients (CV) . Secondly Omega-3- Polyunsaturated fatty acid (PUFA) and tocopherol content (Vit E) in the fresh fish and dried or smoked fish of the highly consumed food fishes would be assessed and the relationship between fish consumption and its PUFA and Vit E content would be known. Also research will focus how lifestyle, socio-demographic factors' influences on the Cardiovascular diseases among community.
2. Justification Since the consumption of marine fish have high omega-3 fatty acid and showed the reduction of death by CVD, there is no record about the content of omega-3 fatty acid in fresh and brackish water fishes and effects on consumption of fresh and brackish water fishes by South Asian population. Nearly 50 % of population of Sri Lankan consume Inland fishes and it is not known the lipids content, omega-3- fatty acids and tocopherol in muscle of these fishes. This would be first study to understand the content of type of lipids , omega-3 fatty acids, tocopherol and the relationship with fish consumption and CVD. This research will identify the formula of cooking and consumption method of fish.
3. Over all Objectives i) Identification of highly consumed food fish varieties (fresh, marine and lagoon) in the district and consumption rate.

   iii) Quantifying the Omega-3 -Polyunsaturated fatty acid and Tocopherol content of flesh of selected highly consumed fishes.

   iv) Compare the lipid profile of the randomly selected CVD patients and apparently healthy subjects and to relate it to PUFAs content of fish v) Assess all the factors related with fish consumption and CVD and to finding a new method of consumption of fish.
4. Literature Review Consumption of fish provides an important nutrient for 135 billions of people worldwide and thus makes a very significant contribution to nutrients (FAO, 2010). Fish consists of polyunsaturated fatty acids in the form of arachidonic acid, eicosapentaenoic acid and docosahexaenoic acid (Kinsella et al.1990). Marine species have high level of PUFAs and those species are less likely consuming by the poor and low income people. And Small pelagic forage fish species have rich PUFAS and they are cheaper and preferably consumed by them (Tacon and Metain, 2009). Increasing consumption of omega-3 fatty acid can benefit health by reducing Cardiovascular diseases (Udani and Ritz, 2013). Kinsella (2005) reported that the increase of unsaturated fatty acids along with the reduction of saturated fats , supports the lowering of blood cholesterol in humans. Din et al., ( 2004) stated that the fish consumption were mainly attributed to the effect of omega-3 polyunsaturated fatty acids which are thought to have several potential cardio protective actions. It was observed that Greenland Eskimos exhibited significantly lower rates of mortality from coronary heart disease (CHD) compared to Danes due to high intake of fish which are rich of omega -3 PUFAs (Menotti et al, 1999 Heidel et al ., 2007). However, Coronary heart disease is still the leading cause of death and disability in the world. Well known risk factors for heart diseases include age, sex, smoking, diet, physical inactivity, high blood pressure, diabetes and high cholesterol level and some more factors associated such as life style, social class, income and occupational factors comprising job stress, combustion products and environmental factors (Yasunori Suematsu et al,2013). The consumption of fish and fish products is recommended as a means of preventing cardiovascular diseases and greatly increased over recent decades in many European countries (Cahu et al .,2004). Modification in the fatty acids profiles by different culinary technologies in cooking fish for consumption alters the nutritive value of final product is major importance of human health. Therefore, the fatty acids profile in fish varied with fresh, processed and cooked form(Garcia-Arias et al., 1998).

   In Sri Lanka, as per the 2011 health ranking report 11.69% of total population death reported due to Coronary heart disease and 7.41% hypertension.Some Nutritionally important fatty acids in seven type of fishes eaten in Sri Lanka has been studied (Liyanage et al., 1989). And the fish consumption behaviors is determined by many factors (Pethiyagoda and Olsen, 2012). . Some nutritionally important fatty acids in seven varieties of fish eaten in Sri Lanka has been studied (Liyanage, et al., 1989) and the fish consumption behaviour is determined by many factors ( Pethiyagoda and Olsen, 2012). The peroximate composition of three species of Scomberoides fish from the Sri Lankan waters was done by (Sutharsiniy and Sivashanthy, 2011b) and stated Scomberoid commonsonianus is good diatetic species. The total lipid and cholesterol content of the five commercial important fish species has been assessed by the ((Sutharsiniy and Sivashanthy, 2011a). Wimalasena and Jayasuriya ( 1996) studied the nutritional analysis of some freshwater fishes in Sri Lanka
5. Methodology 5.1. Study Design Annexure I

   . 5.2.Hypothesis of study Omega-3- fatty acid (PUFAs) and Tocopherol content in fish flesh are high in inland fishes and it prevents CVD diseases as per the interview from the fish eating people.. However, there are many factors such as life style and socio-demographic factors and eating methods of fish will be taken into our study since those are influencing factors of CVD and the Lipid profile of CVD patients and non- CVD people will be compared with fish consumption. This research is justified as a first study in Sri Lanka to understand the relationship of fish consumption and its pattern in naïve and CVD from Eastern Sri Lankan Community 5.3.Study Area

   Study is carried out in Batticaloa District from Vakarai to Kalar.

   5.4. Study Setting

   Study has been planned to collect the information from fish consuming people in the Batticaloa district randomly representing different ethnicity and religion by distributing structured questionnairre.

   5.5. Study Population

   The one fifth (1/5- 2500) of total population in Batticaloa district who consume fish and shellfish as their major proteinous diet will be the subjects of study. In addition, a special focus on the people (250) who have cardiovascular diseases who engaged in treatment.

   5.6. Sampling method

   The selection of subjects for survey will be done by stratified random sampling with consideration of population of divisional secretariat (14) proportionately whole in Batticaloa District. A special focus in the selection of subjects in three DS secretariat ( Manmunai West, KoraliPattu South and Porathivu Pattu).

   Semi-Structured Questionnaire will be used to gather the data with their full permission of subjects.

   Experimental Method- Observation and Analytical Method

   Total fat content and Lipid profile of mostly consuming fishes( muscle) by the subjects ( 10) in fresh , processed and cooked form will be taken for analysis in (triplicates) using standard method. (Annexure2) Omega-3 fatty acids and tocopherol content (triplicates) will be measured from the same set of fishes. Both analytical methods will be carried out in ITI laboratory in Colombo .

   Lipid Profile of Naïve fish consuming people (as control) and People who are suffering CVD diseases will be measured and primary data of demographics, history and lifestyle of the subjects will be studied (. Annexure 2 )

   5.6. Inclusive Criteria People (subjects) must be regular fish consumer and mostly brackish and fresh water consumers.

   5.7. Study Period 3 years study starting from Dec 2013 upto Nov 2016.

   5.8. Materials Used Annexure 2

   5.9. Data Collection

   It will be done by three ways: structured questionnaire, primary data, secondary data, direct interview, Observation data- Market Survey Analytical data- Total lipid content in fish, Fatty acid content in fish, Omega three fatty acid and tocopherol Lipid profile of naïve regular fish consuming people (250) and CVD people who are engaged in treatment .

   Lipid profile for selected subjects (naïve) after 6 month of fish consumption lipid profile will be tested.

   Blood (2ml) will be collected from the subjects for the lipid profile analysis with their consent.

   ( This procedure will be done once the ethical clearance certificate issued)

   5.10 Data Analysis SPSS -19 package , EXCEL and SAS ( if needed) for ranking will be used.

   5.11. Study Sensitization This study will reveal the different fatty acids in fish and the content and these will not be sensitized issue. Since lipid profile of naïve human and CVD people will be treated confidentially and data will be treated same and after research . All data will be destroyed.

   5.12. Consent Statement- Annexure 3

   5.13. Confidentiality Statement Annexure 3

   5.14. Work Plan Annexure 4

   Annexure 2 Phase I This survey will be specially focused on the relationship between consumption of fish /food and its preference of quality, the impact of consumer involvement, role of life styles, experience and habit, quantity intake, time of consumption, socio-demographic characteristics, health and diet beliefs and convenience. It would be done among one in 500 people of total population(525142). That is nearly 1500.

   Of the randomly selected people of fish consumers , nearly 250 people (male & female), aged between 35 to 50 who are engaging in treatment for Cardiac vascular disease (CVD) , hypertension and stroke in three different national hospitals in Eastern Province. The daily fish consumption data, type of fish, amount of fish consumption in three times will be assessed during health survey among patients. During the survey fish eating frequency, cooking method, special ingredients used to cook fish , how many minutes they cooked fish, and processing technique will be interviewed.

   Phase II By doing Market survey (nearly 5 city markets and 5 local markets) the major food fishes would be identified taxonomically and fish consumption rate will be calculated.

   Phase III The total fat content subjected to the study will be extracted according to the Soxhlet protocol (ADAC,1995 ) from the flesh of 10 highly consumed fishes. Total lipid extraction was made with chloroform methanol (2:1) and according to Folich et al ,.(1957) methodology modified by Bligh and Dyer (1959). Fatty acid methyl esters (FAME) will be prepared with methanol using BF3 -MeoH complex, as catalyst, according to the method of Metcalfe et al (1966). Omega-3 fatty acid of the highly consumed fresh, cooked and dried fish muscle would be analyzed using Gas Liquid Chromatography and the tocopherol content will be analyzed using High Performance Liquid Chromatography (HPLC). These would be correlated with consumer preference of fish and CVD. The omega-3 -PUFA and Tocopherol content of all samples would be analyzed at same time. Sample of ten selected highly consumed fish species will be taken for this study. Lipid profile of randomly selected (50) CVD patients who will be selected with the help of the Batticaloa cardiology unit will be taken in our study and it will be monitored monthly for five months.

   Phase IV The correlation between the fish consumption and the cooking methods and life style of the community and Cardiovascular diseases in the Eastern Community will be analyzed.

   Phase V The nutritional composition of identified of selected highly consumed fish and existing cooking method would be studied and new method of cooking style formulated and would be tested and will be introduced among consumers.

ELIGIBILITY:
Inclusion Criteria:

Fish Consumers

Exclusion Criteria:

* Vegetarians

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Effect of fish consumption on Lipid Profiles | 06 months
  Pre and Post interventional lipid profiles were compared with type of fish consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern University, Sri Lanka, Batticaloa, Eastern, Sri Lanka

IPD SHARING:
Plan to Share IPD: No